CLINICAL TRIAL: NCT04765423
Title: [F-18] Fluciclovine (Axumin) PET/CT vs. [F-18] NaF PET/CT in the Evaluation of Prostate Cancer Osseous Metastatic Disease
Brief Title: Fluciclovine (Axumin) PET/CT vs. NaF PET/CT in Prostate Cancer Osseous Metastatic Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE11820
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Malignant Neoplasm of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NaF PET/CT scan and F-18 fluciclovine PET/CT (Experimental): Visit 1: Participant receives a whole body [F-18] NaF PET/CT (diagnostic study)
  Visit 2: Participant receives a whole body [F-18] fluciclovine PET/CT within 3 weeks of Visit 1
  Interventions: Device: [F-18] NaF PET/CT; Device: [F-18] fluciclovine PET/CT

INTERVENTIONS:
Device: [F-18] NaF PET/CT — Radiotracer F-18 NaF used on the PET/CT imaging
Device: [F-18] fluciclovine PET/CT — F-18 fluciclovine (Axumin ®) used on the PET/CT camera
  Other Names: Axumin

SUMMARY:
The purpose of this study is to look at whether F-18 Fluciclovine (i.e. Axumin) is better or as good as F-18 Sodium Fluoride (F-18 NaF) when looking at bone disease from prostate cancer. Axumin is a radioactive agent used on a positron/computed tomography (PET/CT) camera to look for prostate cancer in general.

DETAILED DESCRIPTION:
The study will assess the diagnostic performance of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT as the reference standard. Each bone lesion identified on [F-18] NaF PET/CT will be compared with the level of [F-18] fluciclovine uptake

The primary objective is to assess [F-18] fluciclovine efficacy in the evaluation of osseous metastatic disease in prostate cancer on a lesion-by-lesion comparison with [F-18] NaF as a the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Referred for initial staging or restaging of prostate cancers with clinical suspicion of bone metastases.
* Must understand and voluntarily sign an Informed Consent Document

Exclusion Criteria:

-Cannot tolerate imaging up to 60 minutes of total imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Number of lesions seen by [F-18] NaF PET/CT which are also seen by [F-18] fluciclovine PET/CT | At time of scan, up to 60 minutes per scan
  Agreement of imaging methods as measured by number of lesions seen by [F-18] NaF PET/CT which are also seen by [F-18] fluciclovine PET/CT broken down by diagnostic score on a lesion-by-lesion basis (1 to 5)
  1. Definitely benign
  2. Probably benign
  3. Equivocal
  4. Probably malignant
  5. Definitely malignant
Sensitivity | At time of scan, up to 60 minutes per scan
  Accuracy of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT evaluated via sensitivity
  Sensitivity is the number of true positives (TP) divided by the sum of TP and false negatives (FN):
  Sensitivity = TP / (TP+FN)
Specificity | At time of scan, up to 60 minutes per scan
  Accuracy of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT evaluated via specificity
  Specificity is the number of true Negatives (TN) divided by the sum of TN and false positives (FP):
  Sensitivity = TN / (TN+FP)
Positive Predictive Value (PPV) | At time of scan, up to 60 minutes per scan
  Accuracy of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT evaluated via PPV
  PPV is the number of true TP divided by the sum of TP and FP:
  Sensitivity = TP / (TP+FP)
Negative Predictive Value (NPV) | At time of scan, up to 60 minutes per scan
  Accuracy of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT evaluated via NPV
  NPV is the number of true TN divided by the sum of TN and FN:
  Sensitivity = TN / (TN+FN)
Area under the curve (AUC) | At time of scan, up to 60 minutes per scan
  Accuracy of [F-18] fluciclovine PET/CT compared to [F-18] NaF PET/CT evaluated via AUC using Receiver Operating Characteristic (ROC) curves

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No current plans to share IPD